CLINICAL TRIAL: NCT06306365
Title: Intervention Program on Executive Functions, Participation and Well-being in Older Adults Using Modern Board Games.
Brief Title: Effects of Modern Board Games on Well Being in Older Adults
Acronym: JUMEMO3e+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Miguel de Cervantes (Other)
Collaborators: Centro Doctor Villacián, Valladolid, Spain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI-DOC003-WBOA
Record Dates: First submitted 2024-02-22; First posted 2024-03-12 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-03

CONDITIONS: Executive Functions
Keywords: Modern board game; Executive functions; Social participation; Well-being; Older people

STUDY DESIGN:
Intervention Model Description: A quasi-experimental methodology will be employed, involving both a control group and an experimental group. Randomized control trial.
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Subjects belonging to this group perform a modern board game-based learning.
  Interventions: Behavioral: Modern board game-based learning
- Control (no intervention) (No Intervention): Subjects belonging to this group not perform intervention.

INTERVENTIONS:
Behavioral: Modern board game-based learning — Modern board game-based learning involves using contemporary board games as educational tools. It emphasizes active participation, critical thinking, and social interaction among participants. By integrating strategic thinking and problem-solving within a game context, this approach aims to enhance learning experiences in an engaging and enjoyable manner. In this study, board games have been selected to target and engage executive functions.
  Arms: Experimental

SUMMARY:
The aim of the study is to assess the effects of an intervention using modern board game-based learning in a sample of older individuals. The evaluation will focus on determining if there is a change in executive functions, social participation, and participants' perception of well-being.

DETAILED DESCRIPTION:
The aim of the study is to assess the effects of an intervention using modern board game-based learning in a sample of older individuals. The intervention will last for 12 weeks, incorporating the use of the 16 board games identified in the previous study, which also established the most suitable adaptations and methodologies for this age group. The study will take place in a senior living facility. A quasi-experimental methodology will be employed, involving both a control group and an experimental group. The evaluation will focus on determining if there is a change in executive functions, social participation, and participants' perception of well-being.

ELIGIBILITY:
Inclusion criteria:

* Be residents of the Centro Doctor Villacián (Valladolid).
* Willing to commit to the study.
* Have literacy skills.

Exclusion criteria:

· Presentation of advanced dementia case.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Examination for Mental Disorders of the Elderly | 0 weeks,12 weeks
  The cognitive subscale "CAMCONG" is used, Section B of the CAMDEX-R (Cambridge Examination for Mental Disorders of the Elderly, adapted to Spanish by López-Pousa (2015)). It consists of 60 items (neuropsychological areas). The maximum score is 105 points in this revised option. In the scale validated by López-Pousa and others (1990), the cutoff point that best discriminated between a subject with dementia and one without dementia was 69/70. The scores for the different cognitive functions: orientation (minimun score 0, máximum score 10), language (minimun score 0, maximum score 30), memory (minimum score 0, maximum score 27), attention/calculation (minimum score 0, maximum score 9), praxis (minimun score 0, máximum score 12), abstract thinking (minimum score 0, maximum score 8), perception (mínimum score 0, máximum score 9). Minimum score: 0, total maximum score: 105. Executive function (maximum score is 28). A higher score indicates a better state of executive functions.
Trail Making Test to evaluate Executive Functions | 0 weeks,12 weeks
  As a complement to assess executive functions, the TESEN (Trail Making Test to evaluate Executive Functions) is used, by Portellano Pérez and Martínez Arias (2014). It consists of four subtests (trails) where the evaluated person initiates increasingly complex cognitive processes and demands that measure functions such as working memory, prospective memory, motor processing speed, perceptual speed, inhibition, sustained attention, and alternating attention.
  The TESEN provides three different scores for each trail, which are: execution score (E=hits-errors/time), speed score (V=time in seconds), and accuracy score (P=hits-errors/hits). In the quick correction mode, these values can be converted into decatips, a scale from 1 to 10, where the highest level indicates better development of executive functions.
Assessment of quality of life in older adults and people with disabilities | 0 weeks,12 weeks
  The FUMAT scale (Gómez, Verdugo, Arias, and Navas, 2008) is an assessment instrument composed of 8 subscales that make up Quality of Life. In this study, the dimensions corresponding to will be used: emotional well-being (8 items, minimun score 8, maximum score 32); interpersonal relationships (6 items, minimun score 6, maximum score 24); personal development (8 items, minimum score 8, maximum score 32); social inclusión (9 items, minimun score 9, maximum score 36).
Psychometric development and practical use | 0 weeks,12 weeks
  The Volitional Questionnaire (VQ) by De las Heras, Geist, and Kielhofner (1998) consists of 14 items with a four-level scale, covering the continuum from spontaneous (highest level) to passive (lowest level). The total score of the questionnaire is 56 points and is divided into three scales (exploration, competence, and achievement). A higher score indicates higher levels of volition. Below is indicated the subscale, the number of ítems, the mínimum score and the máximum sore: exploration (5 items, mínimum score 5, maximum score 20), competence (5 items, mínimum score 5, maximum score 20), achievement (4 items, mínimum score 4, maximum score 15).

CONTACTS AND LOCATIONS:
Locations (1):
- European University Miguel of Cervante, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ching-Teng Y. Effect of board game activities on cognitive function improvement among older adults in adult day care centers. Soc Work Health Care. 2019 Oct;58(9):825-838. doi: 10.1080/00981389.2019.1656143. Epub 2019 Aug 21. PMID 31432758
- [Background] Verghese J, Lipton RB, Katz MJ, Hall CB, Derby CA, Kuslansky G, Ambrose AF, Sliwinski M, Buschke H. Leisure activities and the risk of dementia in the elderly. N Engl J Med. 2003 Jun 19;348(25):2508-16. doi: 10.1056/NEJMoa022252. PMID 12815136
- [Background] Estrada-Plana V, Montanera R, Ibarz-Estruga A, March-Llanes J, Vita-Barrull N, Guzman N, Ros-Morente A, Ayesa Arriola R, Moya-Higueras J. Cognitive training with modern board and card games in healthy older adults: two randomized controlled trials. Int J Geriatr Psychiatry. 2021 Jun;36(6):839-850. doi: 10.1002/gps.5484. Epub 2021 Jan 8. PMID 33275804
- [Background] Dartigues JF, Foubert-Samier A, Le Goff M, Viltard M, Amieva H, Orgogozo JM, Barberger-Gateau P, Helmer C. Playing board games, cognitive decline and dementia: a French population-based cohort study. BMJ Open. 2013 Aug 29;3(8):e002998. doi: 10.1136/bmjopen-2013-002998. PMID 23988362
- [Background] Gates NJ, Vernooij RW, Di Nisio M, Karim S, March E, Martinez G, Rutjes AW. Computerised cognitive training for preventing dementia in people with mild cognitive impairment. Cochrane Database Syst Rev. 2019 Mar 13;3(3):CD012279. doi: 10.1002/14651858.CD012279.pub2. PMID 30864747
- [Background] Lee BO, Yao CT, Pan CF. Effectiveness of board game activities for reducing depression among older adults in adult day care centers of Taiwan: a quasi-experimental study. Soc Work Health Care. 2020 Oct-Dec;59(9-10):725-737. doi: 10.1080/00981389.2020.1842576. Epub 2020 Nov 2. PMID 33138738
- [Background] Nakao M. Special series on "effects of board games on health education and promotion" board games as a promising tool for health promotion: a review of recent literature. Biopsychosoc Med. 2019 Feb 19;13:5. doi: 10.1186/s13030-019-0146-3. eCollection 2019. PMID 30820242
- See also: Developing serious games to promote cognitive abilities for the elderly. In 2017 IEEE 5th International Conference on Serious Games and Applications for Health (SeGAH) (pp. 1-8). IEEE. — https://segah.org/2017/docs/Papers/Session%206%20-%20Education/O-S06-4-01.pdf
- See also: Envejecimiento activo: un cambio de paradigma sobre el envejecimiento y la vejez. Aula abierta, 47(1), 45-54. — https://dialnet.unirioja.es/servlet/articulo?codigo=6292831
- See also: Related Info — https://www.who.int/es/news-room/fact-sheets/detail/ageing-and-health